CLINICAL TRIAL: NCT00546715
Title: Placebo-Controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of BMS-790052 in Subjects Chronically Infected With Hepatitis C Virus Genotype 1
Brief Title: A Single Ascending Dose Study of Daclatasvir (BMS-790052) in Hepatitis C Virus Infected Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI444-002
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Panel A (Active Comparator): Daclatasvir - 1 mg
  Placebo - 0 mg
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Dose Panel B (Active Comparator): Daclatasvir - 10 mg
  Placebo - 0 mg
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Dose Panel C (Active Comparator): Daclatasvir - 100 mg
  Placebo - 0 mg
  Interventions: Drug: Daclatasvir; Drug: Placebo
- Dose Panel D (Active Comparator): Daclatasvir - 0.5 - 200 mg (to be determined)
  Placebo - 0 mg
  Interventions: Drug: Daclatasvir; Drug: Placebo

INTERVENTIONS:
Drug: Daclatasvir — Oral Solution, Oral, Single Dose
Drug: Placebo — Oral Solution, Oral, Single Dose

SUMMARY:
The primary purpose of this study is to evaluate the safety profile and tolerability of single oral doses of daclatasvir in subjects with chronic hepatitis C infection

ELIGIBILITY:
Key Inclusion Criteria:

* Chronically infected with hepatitis C virus genotype 1
* Treatment naive or treatment non-responders or treatment intolerant; and not co-infected with HIV or hepatitis B virus
* Hepatitis C virus RNA viral load of ≥ 10*5* IU/mL
* BMI 18 to 35 kg/m²

Key Exclusion Criteria:

* Any significant acute or chronic medical illness which is not stable or is not controlled with medication and not consistent with hepatitis C virus infection
* Major surgery within 4 weeks of study drug administration and any gastrointestinal surgery that could impact the absorption of study drug

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Advanced Clinical Research Institute, Anaheim, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Parexel International Corporation, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Bristol-Myers Squibb Clinical Pharmacology Unit, Hamilton, New Jersey
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University Of Virginia Digestive Health Center Of Excellence, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 centers in United States.
Pre-assignment Details: A total of 95 participants were enrolled, of which 18 received treatment. Remaining 77 participants were not randomized (participants either no longer met study criteria by the time of randomization or were no longer needed as an adequate number of study participants had already been dosed in each dose panel).
Groups:
- Daclatasvir-1 mg: Participants received single dose of daclatasvir 1 mg as oral solution at concentration of 1 mg/mL daily, after fasting for at least 10 hours pre-dose and 4 hours post-dose.
- Daclatasvir-10 mg: Participants received single dose of daclatasvir 10 mg as oral solution at concentration of 1 mg/mL daily, after fasting for at least 10 hours pre-dose and 4 hours post-dose.
- Daclatasvir-100 mg: Participants received single dose of daclatasvir 100 mg as oral solution at concentration of 50 mg/mL daily, after fasting for at least 10 hours pre-dose and 4 hours post-dose.
- Placebo: Participants received single dose of placebo matched to daclatasvir daily, after fasting for at least 10 hours pre-dose and 4 hours post-dose.
Period: Overall Study
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Started | 6 | 5 | 5 | 2
Completed | 6 | 4 | 5 | 2
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed in the safety population defined as all participants who received any study drug treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 5 | 2 | 18
Age, Continuous [Median (Full Range); unit: years] | 43.5 [31 to 48] | 46 [23 to 49] | 44 [32 to 45] | 28 [22 to 34] | 44 [22 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 0 | 8
  Male | 5 | 2 | 1 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs) and Who Died
Description: AEs were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding) or disease which either occurs during study, whether or not related to the study drug. SAEs were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: Day 1 up to Day 7 for non-SAEs and Day 1 to 30 days after study discontinuation for SAEs
Population: Analysis was performed in safety population defined as all participants who received any study drug treatment.
Measure: Number; unit: participants
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 2
participants
  SAEs | 0 | 0 | 0 | 0
  Discontinuations due to AEs | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Sign Measurements and Physical Examination Findings
Description: Participants were assessed by investigator for any clinically significant changes in vital parameters like body temperature, respiratory rate, blood pressure, heart rate and weight. The assessment was performed by a calibrated sphygmomanometer and thermometer for blood pressure and temperature, respectively. Blood pressure and heart rate were measured after at least 5 minutes quiet seating of the subject. Weight was measured at the discharge. The criteria for clinically significant change was as per the investigators discretion.
Time Frame: Day 1 up to Day 7 or Discharge
Population: The analysis was performed in the safety population.
Measure: Number; unit: participants
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 2
participants
  Systolic blood pressure | 0 | 0 | 0 | 0
  Diastolic blood pressure | 0 | 0 | 0 | 0
  Pulse rate | 0 | 0 | 0 | 0
  Respiration rate | 0 | 0 | 0 | 0
  Temperature | 0 | 0 | 0 | 0
  Weight | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Marked Abnormalities in Laboratory Findings
Description: Laboratory marked abnormalities were defined as Hematocrit (low) as <0.85*pre-treatment value, Leukocytes (low) as <0.9*lower limit of normal, Aspartate Aminotransferase (high) as >1.25*upper limit of normal, Creatinine (high) as >1.33*pre-treatment value, Bicarbonate (high) as >1.2*upper limit of normal, Total Protein (high) as >1.1*upper limit of normal, Creatinine Kinase (high) as >1.5*upper limit of normal, Blood in Urine (high) as ≥ 2*upper limit of normal. Participants were fasted for at least 10 hours prior to the collection of blood specimens for clinical laboratory tests.
Time Frame: Day 1 up to Day 7
Population: The analysis was performed in the safety population.
Measure: Number; unit: participants
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 2
participants
  Hematocrit (Low) | 1 | 0 | 0 | 0
  Leukocytes (Low) | 0 | 0 | 1 | 0
  Aspartate Aminotransferase (High) | 1 | 0 | 0 | 0
  Creatinine (High) | 1 | 1 | 1 | 1
  Bicarbonate (High) | 0 | 1 | 0 | 0
  Total Protein (High) | 1 | 0 | 1 | 0
  Creatinine Kinase (High) | 1 | 0 | 0 | 0
  Blood in Urine (High) | 0 | 0 | 1 | 0

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) and Observed Plasma Concentration at 12 Hours (C-12) and 24 Hours (C-24)
Description: Maximum observed plasma concentration following drug administration from the raw plasma concentration-time data. C-12 and C-24 were defined as observed plasma concentration of daclatasvir at 12 hours and 24 hours, respectively. The plasma samples were analyzed for daclatasvir using a validated liquid chromatography-tandem mass spectrometric assay.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 and 72 hours post-dosing on Day 1
Population: The analysis was performed in the pharmacokinetic (PK) set population defined as all participants who received at least single dose of daclatasvir with available valid data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg
Number analyzed (Participants) | 6 | 5 | 5
ng/mL
  Cmax | 15.7 (56) | 177.6 (52) | 2416.5 (27)
  C-12 | 2.7 (49) | 32.2 (28) | 706.7 (51)
  C-24 | 1.1 (65) | 14.2 (44) | 363.2 (55)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-T]), Area Under the Plasma Concentration-time Curve From Time Zero (AUC[INF]) Extrapolated to Infinite Time
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration. It was calculated as the sum of linear trapezoids using non-compartmental analysis. Area under the plasma concentration-time curve from time zero extrapolated to infinite time was estimated as sum of AUC(0-T) and the extrapolated area, computed by the quotient of the last observable concentration and λ, where λ was the slopes of the terminal phases of the plasma concentration-time profiles. The plasma samples were analyzed for daclatasvir using a validated liquid chromatography-tandem mass spectrometric assay.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 and 72 hours post-dosing on Day 1
Population: The analysis was performed in the PK set population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg
Number analyzed (Participants) | 6 | 5 | 5
ng*h/mL
  AUC(0-T) | 126.8 (49) | 1413.9 (45) | 28239.1 (48)
  AUC(0-INF) | 129.1 (49) | 1431.1 (45) | 29256.1 (53)

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax was defined as the time required to reach maximum observed plasma concentration. The plasma samples were analyzed for daclatasvir using a validated liquid chromatography-tandem mass spectrometric assay.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 and 72 hours post-dosing on Day 1
Population: The analysis was performed in the PK set population.
Measure: Median (Full Range); unit: hours
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg
Number analyzed (Participants) | 6 | 5 | 5
hours | 1 [0.5 to 3] | 1 [1 to 1.5] | 1.5 [1 to 3]

7. Secondary Outcome: Plasma Half-life (T-half)
Description: Plasma half-life was defined as the time required for one half of the total amount of administered drug eliminated from the body. The plasma samples were analyzed for daclatasvir using a validated liquid chromatography-tandem mass spectrometric assay.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 and 72 hours post-dosing on Day 1
Population: The analysis was performed in the PK set population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg
Number analyzed (Participants) | 6 | 5 | 5
hours | 9.7 (2.65) | 12.1 (1.97) | 14.0 (6.43)

8. Secondary Outcome: Apparent Total Body Clearance (CLT/F)
Description: Apparent total body clearance (CLT/F) was calculated as Dose/AUC(INF), where CLT was the clearance of the drug and F was the absolute oral bioavailability. The plasma samples were analyzed for daclatasvir using a validated liquid chromatography-tandem mass spectrometric assay.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 and 72 hours post-dosing on Day 1
Population: The analysis was performed in the PK set population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg
Number analyzed (Participants) | 6 | 5 | 5
mL/min | 129.1 (48) | 116.5 (43) | 57.0 (49)

9. Secondary Outcome: Decline From Baseline in log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: The Roche TaqMan HCV quantitative assay was used for analysis with detection limit of 10 IU/mL. Positive value indicated reduction from baseline in HCV RNA while negative value indicated an increase from baseline in HCV RNA. Baseline HCV RNA was defined as the pre-dose value on Day 1 log10 HCV RNA.
Time Frame: Pre-dose, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 144 hours post-dose on Day 1
Population: The analysis was performed in the pharmacodynamic (PD) population defined as participants who received at least one dose of study medication with available valid data.
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 2
log IU/mL
  Decline From Baseline to 24 hours | 2.12 (0.57) | 3.24 (0.51) | 3.28 (0.35) | -0.12 (0.29)
  Maximum Decline | 2.44 (0.80) | 3.12 (0.66) | 4.06 (0.53) | 0.06 (0.11)

10. Secondary Outcome: Time to Reach Maximum Decline in Plasma Hepatitis C Virus RNA Levels From Baseline
Description: Participants were assessed for time to reach maximum decrease in log10 hepatitis C virus RNA level. Baseline HCV RNA was defined as the pre-dose value on Day 1 log10 HCV RNA.
Time Frame: Pre-dose, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 144 hours post-dose on Day 1
Population: The analysis was performed in the PD population defined as participants who received at least one dose of study medication with available valid data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 2
hours | 16.4 (7.8) | 43.2 (56.74) | 105.60 (55.25) | 144 (0)

11. Secondary Outcome: Change From Baseline in Heart Rate to Day 7 or Discharge
Description: Changes in heart rate from baseline were measured after the participants were supine for at least 5 minutes. Baseline was defined as the Day 1 pre-dose measurement. The normal heart rate lies between 60-90 beats per minute (bpm), below 60 bpm and above 90 bpm were considered as bradycardia and tachycardia, respectively.
Time Frame: Baseline (Day 1), Day 7 or Discharge
Population: The analysis was performed in the safety population.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 2
bpm | 7.3 (16.2) | 7.6 (9.3) | 1.6 (8.5) | 14 (1.4)

12. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters (PR, QRS, QT, and QTc Intervals) to Day 7 or Discharge
Description: The ECG was recorded after the participant was in a supine position for at least 5 minutes. Baseline was defined as the Day 1 pre-dose measurement. The PR interval was defined as the beginning of the P wave to the beginning of the QRS complex, and represents the time taken by electrical impulse to travel from the sinus node through the atrioventricular (AV) node. The QRS complex represented the rapid depolarization of the right and left ventricles. The QT interval was defined as the time from the start of the Q wave to the end of the T wave, and represents the time taken for ventricular depolarization and repolarization. QTc was defined as corrected QT interval at a heart rate of 60 bpm. QTc was estimated using Bazett's formula and Fredericia's formula.
Time Frame: Baseline (Day 1), Day 7 or Discharge
Population: The analysis was performed in the safety population.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 2
msec
  QT Interval | -27.5 (32.7) | -18.6 (29.2) | -1.2 (27.8) | -36 (14.1)
  QTc Fridericia Interval | -13.3 (10.5) | -5.6 (14.7) | 0.4 (11.4) | -12.5 (19.1)
  QTc Bazett Interval | -5.5 (21.0) | 1.2 (12.7) | 1.8 (7.2) | 1 (21.2)
  QRS Width | -2.3 (4.7) | 1 (11.3) | -3.6 (8.2) | 0 (0)
  PR Interval | -6.7 (9.9) | 2.4 (10.3) | -4.4 (11.2) | -7 (7.1)

13. Secondary Outcome: Change From Baseline in Blood Pressure to Day 7 or Discharge
Description: Changes in blood pressure from baseline were measured after the participants were supine for at least 5 minutes. Baseline was defined as the Day 1 pre-dose measurement.
Time Frame: Baseline (Day 1), Day 7 or Discharge
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Number analyzed (Participants) | 5 | 4 | 3 | 1
mmHg
  Diastolic blood pressure | 9.6 (7.3) | 4.3 (5.9) | 3.7 (12.7) | 1 (NA) — Only 1 participant was available for assessment, hence value of standard deviation is not applicable.
  Systolic blood pressure | 14 (4.4) | 1 (15.7) | 6 (17.5) | -2 (NA) — Only 1 participant was available for assessment, hence value of standard deviation is not applicable.

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 7 (for non-SAEs), Day 1 to 30 days after study discontinuation (for SAEs)
Description: On-treatment period
Arm/Group | Daclatasvir-1 mg | Daclatasvir-10 mg | Daclatasvir-100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 3/6 | 3/5 | 1/5 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir-1 mg (N=6) | Daclatasvir-10 mg (N=5) | Daclatasvir-100 mg (N=5) | Placebo (N=2)
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.